CLINICAL TRIAL: NCT06825754
Title: The Value of Serum MicroRNA-21-5p and LncRNAgadd7 Expression Levels in Predicting the Severity and Prognosis of ARDS ( Acute Respiratory Distress Syndrome )
Status: Completed | Type: Observational
Sponsor: Shao Yuekai (Other)
Responsible Party: Sponsor-Investigator, Shao Yuekai, Researcher, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Other Study IDs: KLLY-2023--198
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survival Group
- Death Group

SUMMARY:
By measuring the expression levels of MicroRNA-21-5p (miR-21-5p) and LncRNAgadd7 in the peripheral blood of ARDS patients, the study aims to explore the correlation between these levels and the severity and prognosis of ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Meets the Berlin Criteria for ARDS;
3. Diagnosed with ARDS within 48 hours;
4. Signed informed consent.

Exclusion Criteria:

1. Immunosuppressed patients: including those on immunosuppressive drugs, history of stem cell transplantation, etc.;
2. Patients with malignant tumors;
3. Pregnant women;
4. Patients discharged from the ICU within 48 hours;
5. History of chronic lung diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS ( Acute Respiratory Distress Syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
The expression levels of MicroRNA-21-5p (miR-21-5p) | 28 days
the expression levels of LncRNAgadd7 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China